CLINICAL TRIAL: NCT01340820
Title: A Phase 1, Randomized, Controlled, Double-blind, Dose-Escalation Study to Evaluate the Safety and Immunogenicity of AERAS-422 in Healthy Adults
Brief Title: Study of AERAS 422 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aeras (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-007-422
Record Dates: First submitted 2011-02-24; First posted 2011-04-25 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — BCG Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AERAS-422 Low dose (Experimental): >=10^5 to < 10^6 CFU
  Interventions: Drug: AERAS-422
- AERAS-422 High Dose (Experimental): >=10^6 CFU
  Interventions: Drug: AERAS-422
- BCG Tice (Active Comparator): BCG Tice 1-8 x 10^5 CFU
  Interventions: Drug: BCG Tice

INTERVENTIONS:
Drug: AERAS-422 — rBCG
  Other Names: BCG Tice
  Arms: AERAS-422 High Dose; AERAS-422 Low dose
Drug: BCG Tice — 1-8 x 10^5 CFU
  Arms: BCG Tice

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of AERAS-422 in healthy, BCG-naïve adults.

DETAILED DESCRIPTION:
This is a Phase I, randomized, controlled, double-blind, dose-escalation study of AERAS-422. This study will be conducted in 24 HIV-negative, healthy adults who are BCG-naïve and negative for prior exposure to Mtb at enrollment. The study will be conducted at one or more clinical research sites in the United States.

AERAS-422 will be administered on Study Day 0 as a single 0.1 mL intradermal (ID) injection containing either >= 10^5 to <10^6 CFU (low-dose) or >=10^6 CFU (high-dose). BCG Tice® will be used as an active control for AERAS-422 and will be administered as a single 0.1 mL ID injection containing 1-8 x 10^5 CFU on Study Day 0.

ELIGIBILITY:
Inclusion Criteria:

-≥18 years and ≤45 years of age on randomization day

* Has general good health, confirmed by medical history and physical examination
* Has a screening body mass index (BMI) ≥19 and <33
* Females physically capable of pregnancy (not sterilized and still menstruating or within 1 year of the last menses if menopausal) in sexual relationships with men must use acceptable method of avoiding pregnancy from 28 days prior to randomization through the end of the study.
* Acceptable methods of avoiding pregnancy -Females physically capable of pregnancy must have:
* Negative urine pregnancy test within 21 days prior to randomization AND within 24 hours prior to Study Day 0 vaccination
* Ability to complete all protocol study visits and be reachable by telephone
* Provided written informed consent prior to screening evaluations
* Completed simultaneous enrollment in the Aeras Vaccine Registry protocol

Exclusion Criteria:

* Acute illness on randomization day
* Oral temperature >=37.5 degrees C on randomization day
* Abnormal laboratory values from blood collected within 21 days prior to randomization as follows:
* Positive test for hepatitis B core antibody or hepatitis C antibody
* Positive test for HIV
* Positive urine test for opiates, cocaine, or amphetamines
* Positive QuantiFERON®-TB Gold test
* History of treatment for active or latent tuberculosis infection
* Other evidence of active or latent tuberculosis, in the opinion of the investigator
* Tuberculin skin test (TST) within 90 days prior to randomization
* History or evidence of allergic disease or reaction that in the opinion of the investigator is likely to be exacerbated by any component of AERAS-422 or BCG Tice
* History or evidence of autoimmune disease, immunosuppression, or immunodeficiency, in the opinion of the investigator
* History or evidence of cheloid formation, axillary or cervical lymphadenopathy, or other dermatologic or anatomic findings that, in the opinion of the investigator, may interfere with the assessment of injection site reactions
* History or evidence of any other acute or chronic disease or condition that, in the opinion of the investigator, may compromise the safety of the subject or interfere with the evaluation of the vaccine safety or immunogenicity
* Medical, psychiatric, occupational, or substance abuse problems that, in the opinion of the investigator, will make it unlikely the subject will comply with the protocol
* Inability to discontinue daily prescription medications (except contraceptives) during the study.
* Received immunosuppressive medication within 45 days prior to randomization (inhaled and topical corticosteroids are permitted)
* Received investigational drugs or vaccine products within 182 days prior to randomization, or planned participation in any other investigational study during the study
* Received investigational Mtb vaccine at any time prior to randomization
* Received vaccination or immunotherapy with a BCG product at any time prior to randomization
* Received immunoglobulin or blood products within 45 days prior to randomization
* Received inactivated influenza vaccine within 14 days prior to randomization or any other standard vaccine within 45 days prior to randomization.
* Received systemic antibiotics within 14 days prior to randomization

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-12; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Safety | Days 0, 3, 7, 14, 28, 56, 84, 112, 140 & 182
  Assessment of collected unsolicited and solicited adverse events (including site of injection reaction (pain, erythema, induration, ulceration, drainage, and scarring), regional lymphadenopathy (axillary and cervical), fever, headache, myalgia, arthralgia and fatigue. The adverse event collection timeframe includes all events that occur up to 56 days after study vaccination. Assessment of serious adverse events will be based on events collected throughout the duration of the study. All safety data will be evaluated before moving into the next successive dose level.

SECONDARY OUTCOMES:
Immunogenicity | Days 0, 14, 28, 56, 84, 112, 140 and 182
  Measurement of immunogenicity based on the percentage of cytokine producing T cells.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hoft, MD, Principal Investigator — St. Louis University Hospital
Locations (1):
- St. Louis University Hospital, St Louis, Missouri, United States

REFERENCES:
- [Derived] Hoft DF, Blazevic A, Selimovic A, Turan A, Tennant J, Abate G, Fulkerson J, Zak DE, Walker R, McClain B, Sadoff J, Scott J, Shepherd B, Ishmukhamedov J, Hokey DA, Dheenadhayalan V, Shankar S, Amon L, Navarro G, Podyminogin R, Aderem A, Barker L, Brennan M, Wallis RS, Gershon AA, Gershon MD, Steinberg S. Safety and Immunogenicity of the Recombinant BCG Vaccine AERAS-422 in Healthy BCG-naive Adults: A Randomized, Active-controlled, First-in-human Phase 1 Trial. EBioMedicine. 2016 May;7:278-86. doi: 10.1016/j.ebiom.2016.04.010. Epub 2016 Apr 19. PMID 27322481